CLINICAL TRIAL: NCT07006090
Title: A Prospective, Observational, Post-Market Registry to Collect Real-World Clinical Data on the Use of the Histolog Scanner in Multiple Disease Areas.
Brief Title: EU Post-Market Registry to Collect Real-World Clinical Data on the Use of the Histolog Scanner.
Acronym: EU - ORCHID
Status: Not yet recruiting | Type: Observational
Sponsor: SamanTree Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: ORCHID Histolog Registry - EU
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Adult Patients Undergoing a Surgery or a Medical Procedure With Use of Histolog® Scanner; Whatever the Disease Area
Keywords: Histolog Scanner

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Adult patients undergoing a surgery or a medical procedure with use of Histolog® Scanner: unique cohort in the study
  Interventions: Device: Histolog Scanner

INTERVENTIONS:
Device: Histolog Scanner — Histolog Scanner intended to allow imaging of the internal microstructure of tissues including, but not limited to, the identification of cells, vessels and their organization or architecture.

SUMMARY:
The goal of this observational study is to gather real-world evidence on the performance and safety of the Histolog® Scanner (HLS) when used as intended. HLS is a real-time ex-vivo tissue imaging device.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old at the time of consenting
* Undergoing a surgery or a medical procedure with use of Histolog® Scanner
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Active participation in a drug, device, or other medical intervention study that has not reached its primary endpoint at the time of consenting
* Patients under judicial protection, legal guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients undergoing a surgery or a medical procedure with use of Histolog Scanner.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2034-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Number of confirmed medical interventions based on Histolog® image readings. | From enrolment to diagnosis confirmation at post surgery follow-up visit (V2: 37 days after enrolment)

SECONDARY OUTCOMES:
Concordance between the assessment of Histolog® images and the final pathology assessment expressed as sensitivity, specificity, positive predictive value, and negative predictive value | From enrolment to post surgery follow-up visit (V2: 37 days after enrolment)
Re-operation rates if Histolog® used for intra-operative assessment | From surgery (V1: Day 0) to post surgery follow-up visit (V2: +30 days)
Cancer-free survival up to 5 years of follow-up | From enrolment to the end of 5 years follow-up
Evaluation of usage patterns across different indications and application profiles. | From enrolment to the end of 5 years follow-up.
Device deficiency defined as any inadequacy in the identity, quality, durability, reliability, safety or performance of a device, including malfunction, use errors or inadequacy in information supplied by the manufacturer. | From first patient surgery visit (V1: Day 0) to last patient surgery visit.

IPD SHARING:
Plan to Share IPD: No